CLINICAL TRIAL: NCT00289536
Title: Advate Antihemophilic Factor (Recombinant), Plasma/Albumin-Free Method (ADVATE rAHF-PFM): A Phase 4 Study to Determine the Pharmacokinetic Response of Patients Diagnosed With Severe Hemophilia A to Different Doses of ADVATE rAHF-PFM
Brief Title: Dose-Response Study of Recombinant Factor VIII Manufactured Protein-Free (rAHF-PFM) in Patients With Hemophilia A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 060403
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose (Experimental)
  Interventions: Biological: Antihemophilic factor, recombinant, manufactured protein-free
- Medium Dose (Experimental)
  Interventions: Biological: Antihemophilic factor, recombinant, manufactured protein-free
- High Dose (Experimental)
  Interventions: Biological: Antihemophilic factor, recombinant, manufactured protein-free

INTERVENTIONS:
Biological: Antihemophilic factor, recombinant, manufactured protein-free — 15 IU/kg rAHF-PFM
  Arms: Low Dose
Biological: Antihemophilic factor, recombinant, manufactured protein-free — 30 IU/kg rAHF-PFM
  Arms: Medium Dose
Biological: Antihemophilic factor, recombinant, manufactured protein-free — 50 IU/kg rAHF-PFM
  Arms: High Dose

SUMMARY:
The purpose of this study is to determine the effect of 3 doses of ADVATE rAHF-PFM on initial recovery (% increase [IU/dL] per IU/kg infused) and major single-infusion pharmacokinetic parameters. The 3 doses are 15, 30, and 50 IU/kg. Prior to each infusion, subjects will not have received treatment with a factor VIII concentrate for at least 3 days. Blood samples will be drawn within 30 minutes pre-infusion and at 0.25, 0.5, 1, 3, 6, 9, 24, 28, 32 and 48 hours post-infusion. A washout period of at least 3 days, but no more than 30 days between the last blood draw and the next infusion will be observed. During participation, subjects will maintain their preexisting treatment regimens with ADVATE rAHF-PFM or other factor VIII concentrate.

A secondary objective is to investigate the relationship between pharmacokinetic parameters at each dose level and the levels of von Willebrand factor ristocetin cofactor activity and von Willebrand factor antigen at baseline.

ELIGIBILITY:
Inclusion Criteria:

* The subject has severe hemophilia A as defined by a baseline factor VIII activity <1% of normal; tested at screening. (A minimum washout period of 3 days is required before the blood sample can be drawn to determine baseline factor VIII levels.)
* The subject has a documented history of at least 150 exposure days to factor VIII concentrates (either plasma-derived or recombinant).
* The subject is within 12 to 65 years of age.
* The subject has a Karnofsky performance score >60.
* The subject is human immunodeficiency virus negative (HIV-) or HIV+ with CD4 count >=400 cells/mm3 (CD4 count determined at screening, if necessary).
* The subject or subject´s legally authorized representative has provided written informed consent.

Exclusion Criteria:

* The subject has a known hypersensitivity to mouse or hamster proteins or to factor VIII concentrates.
* The subject has a history of factor VIII inhibitors with titer >=0.8 BU (Bethesda Assay) or >=0.4 BU (Nijmegen modification of the Bethesda Assay) any time prior to screening.
* The subject has a detectable factor VIII inhibitor at screening, >=0.4 BU (Nijmegen modification of the Bethesda Assay), in the Baxter central laboratory.
* The subject has severe chronic liver disease as evidenced by, but not limited to, any of the following: International Normalized Ratio (INR) >1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices.
* The subject has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (e.g. qualitative platelet defect or von Willebrand´s Disease).
* The subject has participated in another investigational study within 30 days of enrollment.
* The subject´s clinical condition may require a major or moderate surgery (estimated blood loss >500 mL) during the period of participation in the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-02-02 (Actual); Primary Completion 2007-04-01 (Actual); Study Completion 2007-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- United States (8):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Peoria, Illinois
  - Iowa City, Iowa
  - New Brunswick, New Jersey
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted in the United States at 8 study sites.
Pre-assignment Details: Participants were screened for a maximum of 30 days. Participants were randomized to a single sequence of the 3 doses of Antihemophilic Factor (Recombinant), Plasma/Albumin-Free Method (rAHF-PFM). Before each pharmacokinetic evaluation, at least a 3 day washout period and negative factor VIII inhibitor titer was required.
Groups:
- Low Dose: 15 IU/kg rAHF-PFM
- Medium Dose: 30 IU/kg rAHF-PFM
- High Dose: 50 IU/kg rAHF-PFM
Period: Period 1
Arm/Group | Low Dose | Medium Dose | High Dose
Started | 9 | 8 | 9
Completed | 9 | 8 | 9
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Low Dose | Medium Dose | High Dose
Started | 10 (5 participants received Medium Dose and 5 participants received High Dose in Period 1) | 9 (5 participants received Low Dose and 4 participants received High Dose in Period 1) | 7 (4 participants received Low Dose and 3 participants received Medium Dose in Period 1)
Completed | 10 | 9 | 7
Not Completed | 0 | 0 | 0
Period: Period 3
Arm/Group | Low Dose | Medium Dose | High Dose
Started | 7 (3 participants received Medium Dose and 4 participants received High Dose in Period 2) | 9 (5 participants received Low Dose and 4 participants received High Dose in Period 2) | 10 (5 participants received Low Dose and 5 participants received Medium Dose in Period 2)
Completed | 7 | 9 | 9
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treated Participants: Participants who received at least 1 infusion of rAHF-PFM.
Arm/Group | Treated Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Initial Recovery
Description: Percent increase in factor VIII concentration per dose from pre- to post-infusion
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion to 30 minutes post-infusion
Population: Per protocol population: participants who were randomized, received all 3 doses of rAHF-PFM, and had pharmacokinetic assessments.
Measure: Median (Full Range); unit: IU/dL per IU/kg
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
IU/dL per IU/kg | 1.7 [0.5 to 2.7] | 1.6 [0.4 to 2.6] | 1.8 [1.2 to 2.8]
Statistical Analysis 1: Comparison: Low Dose vs Medium Dose vs High Dose; Null Hypothesis: The mean log initial recovery will be the same in each dose group; Test type: Superiority or Other; p = 0.1662, ANOVA; Repeated measures ANOVA with dose as fixed effect

2. Secondary Outcome: Area Under the Curve/Dose
Description: Area under the plasma factor VIII concentration versus time curve (AUC) estimated by linear trapezoidal method per dose.
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: IU*hour/dL per IU/kg
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
IU*hour/dL per IU/kg | 21.2 [8.8 to 43.3] | 20.5 [6.5 to 42.2] | 22.3 [14.5 to 46.9]
Statistical Analysis 1: Comparison: Low Dose vs Medium Dose vs High Dose; Null Hypothesis: The mean log AUC/dose will be the same in each dose group; Test type: Superiority or Other; p = 0.0965, ANOVA — No adjustments were made for multiple comparisons; Repeated measures ANOVA with dose as fixed effect

3. Secondary Outcome: Terminal Half-life
Description: Computed from the regression slope in the terminal phase of the model (the slope is biphasic). Terminal half life is the time it takes for the plasma concentration or the amount of drug in the body to be reduced by 50%.
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
hour | 11.3 [5.4 to 19.9] | 12.3 [6.0 to 20.0] | 11.2 [7.5 to 25.1]
Statistical Analysis 1: Comparison: Low Dose vs Medium Dose vs High Dose; Null Hypothesis: The mean terminal half-life will be the same in each dose group; Test type: Superiority or Other; p = 0.5057, ANOVA; Repeated measures ANOVA with dose as fixed effect

4. Secondary Outcome: Area Under the Curve
Description: AUC estimated by linear trapezoidal method. The linear trapezoidal method is a numerical method used to approximate the area under a curve.
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: IU*hour/dL
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
IU*hour/dL | 300.1 [124.5 to 544.9] | 595.2 [167.8 to 1104.8] | 1055.8 [712.1 to 1778.3]

5. Secondary Outcome: Total Area Under the Curve
Description: Total AUC with extrapolation using the slope of the β-phase
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: IU*hour/dL
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
IU*hour/dL | 318.5 [131.8 to 648.8] | 616.3 [194.4 to 1264.8] | 1116.0 [723.3 to 2344.9]

6. Secondary Outcome: Total Area Under the Moment Curve
Description: Total area under the first moment curve (AUMC) estimated by linear trapezoidal methods
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: IU*hour^2/dL
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
IU*hour^2/dL | 4760.9 [1042.9 to 16315.9] | 7115.1 [2673.6 to 28374.2] | 16464.7 [7111.4 to 77439.7]

7. Secondary Outcome: Weight-adjusted Clearance
Description: Computed as weight-adjusted dose divided by total AUC
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: mL/kg*hour
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
mL/kg*hour | 4.71 [2.34 to 11.38] | 4.88 [2.37 to 15.43] | 4.47 [2.13 to 6.91]

8. Secondary Outcome: Mean Residence Time
Description: Computed as total AUMC divided by total AUC
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
hour | 14.6 [7.2 to 25.1] | 12.8 [7.5 to 24.7] | 14.7 [9.2 to 33.0]

9. Secondary Outcome: Volume of Distribution at Steady State
Description: Computed as weight-adjusted CL * Mean Residence Time
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: dL/kg
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
dL/kg | 0.7 [0.4 to 0.9] | 0.6 [0.4 to 3.4] | 0.6 [0.3 to 0.8]

10. Secondary Outcome: Maximum Plasma Concentration
Description: Maximal factor VIII concentration after infusion
Time Frame: Pharmacokinetic evaluations: 30 minutes pre-infusion up to 48 hours post-infusion
Population: as for outcome 1
Measure: Median (Full Range); unit: IU/dL
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 23 | 23 | 23
IU/dL | 26.0 [13.0 to 42.0] | 50.0 [14.0 to 79.0] | 93.0 [65.0 to 143.0]

11. Secondary Outcome: Pre-infusion Von Willebrand Factor Ristocetin Cofactor Activity (VWF:Rco)
Description: Percentage of normal VWF:Rco activity. Normal is a lab standard consisting of a non-hemophilic population. Relationships between baseline VWF:Rco and pharmacokinetic parameters (initial recovery, total AUC/dose, and half-life) were evaluated statistically.
Time Frame: At baseline and before each pharmacokinetic evaluation
Population: Intent to treat: participants who received at least 1 of the 3 infusions of rAHF-PFM and had pharmacokinetic evaluation(s)
Measure: Median (Full Range); unit: Percent of normal VWF:Rco activity
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 26 | 26 | 26
Percent of normal VWF:Rco activity | 83.0 [40 to 152] | 80.5 [49 to 186] | 80.5 [33 to 182]
Statistical Analysis 1: Comparison: Low Dose vs Medium Dose vs High Dose; Regression analysis: Relationship of initial recovery to pre-infusion level of VWF:Rco with dose groups combined; Test type: Superiority or Other; p = 0.7048, Regression, Linear — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Low Dose vs Medium Dose vs High Dose; Regression analysis: relationship of AUC/Dose to pre-infusion level of VWF:Rco with dose groups combined; Test type: Superiority or Other; p = .0322, Regression, Linear — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: Low Dose vs Medium Dose vs High Dose; Regression analysis: relationship of terminal half-life to pre-infusion level of VWF:Rco with dose groups combined; Test type: Superiority or Other; p = 0.0056, Regression, Linear — No adjustments were made for multiple comparisons

12. Secondary Outcome: Pre-infusion Von Willebrand Factor Antigen (VWF:Ag)
Description: Percentage of VWF:Ag. Relationships between baseline VWF:Ag and pharmacokinetic parameters (initial recovery, total AUC/dose, and half-life) were evaluated statistically.
Time Frame: At baseline and before each pharmacokinetic evaluation
Population: as for outcome 11
Measure: Median (Full Range); unit: U/dL
Arm/Group | Low Dose | Medium Dose | High Dose
Number analyzed (Participants) | 25 | 26 | 26
U/dL | 103.0 [57 to 307] | 117.0 [63 to 309] | 109.5 [61 to 329]
Statistical Analysis 1: Comparison: Low Dose vs Medium Dose vs High Dose; Regression analysis: relationship of initial recovery to pre-infusion level of VWF:Ag with dose groups combined; Test type: Superiority or Other; p = 0.3696, Regression, Linear — No adjustments were made for multiple comparisons
Statistical Analysis 2: Comparison: Low Dose vs Medium Dose vs High Dose; Regression analysis: relationship of AUC/Dose to pre-infusion level of VWF:Ag with dose groups combined; Test type: Superiority or Other; p = 0.0001, Regression, Linear — No adjustments were made for multiple comparisons
Statistical Analysis 3: Comparison: Low Dose vs Medium Dose vs High Dose; Regression analysis: relationship of terminal half-life to pre-infusion level of VWF:Ag with dose groups combined; Test type: Superiority or Other; p < 0.0001, Regression, Linear — No adjustments were made for multiple comparisons

ADVERSE EVENTS:
Time Frame: 15 months
Description: AEs were collected by the investigators at study visits, and may result from laboratory and vital sign assessments collected or measured at the study visits
Groups:
- Safety Population (26 Participants): Participants who received at least 1 infusion of rAHF-PFM
Arm/Group | Safety Population (26 Participants)
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 4/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (26 Participants) (N=26)
Headache (Nervous system disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs vary per individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥45 days prior to submission or communication. Baxter may request an additional delay of up to 60 days (e.g., to allow for intellectual property protection).